CLINICAL TRIAL: NCT00483639
Title: Social Anxiety and Avoidance in Head and Neck Cancer Patients
Brief Title: Study of Anxiety and Avoidance of Others in Patients Previously Treated for Head and Neck Cancer
Status: Completed | Type: Observational
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Kirsten Haman, PhD, Research Assistant Professor; Psychologist, Vanderbilt-Ingram Cancer Center
Other Study IDs: VICC HN 0397; VU-VICC-HN-0397; VU-VICC-IRB-030785
Record Dates: First submitted 2007-06-06; First posted 2007-06-07 (Estimated); Last update posted 2013-03-15 (Estimated); Status verified 2013-03

CONDITIONS: Anxiety Disorder; Head and Neck Cancer; Lung Cancer
Keywords: anxiety disorder; long-term effects secondary to cancer therapy in adults; head and neck cancer; non-small cell lung cancer; small cell lung cancer
MeSH Terms: conditions — Anxiety Disorders; Head and Neck Neoplasms; Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma | interventions — Psychiatric Rehabilitation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Medical chart review — medical chart review
Other: Liebowitz Social Anxiety Scale and the Social Phobia and Anxiety Inventory — survey administration
  Other Names: survey administration
Procedure: management of therapy complications — management of therapy complications
Procedure: Structured Clinical Interview for the Diagnostic and Statistical Manual-IV SCID — psychosocial assessment
  Other Names: psychosocial assessment
Other: Functional Assessment of Cancer Therapy-General (FACT-G) — survey administration

SUMMARY:
RATIONALE: Patients who undergo treatment for head and neck cancer may become anxious and avoid contact with other people. Learning how cancer treatment may cause anxiety in patients with head and neck cancer may help improve the quality of life in these patients.

PURPOSE: This clinical trial is studying anxiety and avoidance of others in patients previously treated for head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the relationship between treatment-provoked social anxiety and avoidance in patients previously treated for head and neck cancer.
* Determine the relationship between pre-cancer psychiatric diagnosis and post-treatment social anxiety and avoidance in these patients.
* Determine the effect of social anxiety and/or avoidance on the quality of life of these patients.
* Investigate the specificity of these relationships in patients with head and neck cancer by comparing patients with head and neck cancer to patients with lung cancer.

OUTLINE: This is a cross-sectional study. Patients are stratified according to prior treatment type (significantly impairing [surgery] vs less impairing [chemotherapy/radiotherapy]).

Patients undergo a face-to-face interview with a mental health clinician over 2 hours. Patients complete multiple psychiatric/psychological assessments during the interview, including the Structured Clinical Interview for DSM-IV (SCID); the Liebowitz Social Anxiety Scale (SAS); the Performance Status Scale for Head and Neck Cancer Patients (PSS-HN); the Social Phobia and Anxiety Inventory (SPAI); the State-Trait Anxiety Inventory (STAI); Response to Stress Questionnaire, Cancer Version (RSQ-CV); the Functional Assessment of Cancer Therapy (FACT-HNC (head neck cancer) or LC); the Voice Handicap Index (VHI); and the Body Image Scale (BIS).

Cancer treatment and medical history information are gathered from patients' medical records.

ELIGIBILITY:
PATIENT CHARACTERISTICS:

* Diagnosis of 1 of the following:

  * Head and neck cancer
  * Lung cancer (control group)
* Must have received treatment for head and neck cancer or lung cancer within the past 5 years

PATIENT CHARACTERISTICS:

* Able to speak and read English to answer surveys, interviews, and questionnaires

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People who have been treated for head and neck cancer.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2003-11; Primary Completion 2006-03 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Level of social anxiety and avoidance in HNC patients post-treatment | at study entry, day 1
  Measured by the Liebowitz Social Anxiety Scale and the Social Phobia and Anxiety Inventory, containing 24 items with each item separately rated for fear as 0 (none), 1 (mild), 2 (moderate) to 3 (severe)and for avoidance behavior as 0 (never), 1 (occasionally), 2 (often), to 3 (usually). Scores are summed with lower values indicating lower levels of social anxiety and avoidance.

SECONDARY OUTCOMES:
Relationship between pre-cancer psychiatric diagnosis and post-treatment social anxiety and avoidance | at study entry
  Assessed using the Structured Clinical Interview for the Diagnostic and Statistical Manual-IV SCID lifetime diagnostic status (pre-cancer diagnosis) and related to the outcome for social anxiety measures. The SCID does not involve a specific scoring of responses. Trained interviewers ask questions that may involve yes/no answers or more detailed explanations. They make their diagnoses based on their experience and training. For this outcome, interviews results will be compared to and contrasted with scores on the Liebowitz Social Anxiety Scale and Social Phobia and Anxiety Inventory.
Quality of Life | at study entry, day 1
  Each patient is scored on the Functional Assessment of Cancer Therapy-General (FACT-G) with 4 related sub-scales (physical, social/family, emotional, functional well-being. To generate sub-scale scores, physical and emotional items are reverse coded and items are then summed, such that higher values indicate better quality of life. Thus, each sub-scale score ranges from 0 (not at all, worse outcome) to 4 (very much, better outcome) with a minimum total score of 0 (worst quality of life) to a maximum of 16 (good quality of life).
Comparison of social anxiety and avoidance in patients with head and neck cancer to patients with lung cancer | at study entry, day 1
  Measured by the Liebowitz Social Anxiety Scale and the Social Phobia and Anxiety Inventory, containing 24 items with each item separately rated for fear as 0 (none), 1 (mild), 2 (moderate) to 3 (severe)and for avoidance behavior as 0 (never), 1 (occasionally), 2 (often), to 3 (usually). Scores are summed with lower values indicating lower levels of social anxiety and avoidance. Scores in study participants will be compared to scores in studies of social anxiety and avoidance in lung cancer patients

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Haman, PhD, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (2):
- United States (2):
  - MBCCOP - Meharry Medical College - Nashville, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee